CLINICAL TRIAL: NCT06633406
Title: Intelligence and Neurodevelopmental Disorders After Prenatal Exposure to General Anaesthesia for Maternal Abdominal Surgery: A Propensity Score Weighted Multicentre Clinical Bidirectional Cohort Study.
Brief Title: Intelligence and Neurodevelopmental Disorders After Prenatal Exposure to General Anaesthesia
Acronym: PAE-IQ
Status: Enrolling by invitation | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S68647
Record Dates: First submitted 2024-09-20; First posted 2024-10-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: General Anaesthesia During Pregnancy
Keywords: anaesthesia; anaesthesia-induced neurotoxicity; pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prenatal Anaesthesia Exposure: Children exposed in utero to maternal general anaesthesia to allow laparoscopy or laparotomy for appendicectomy, adnexal pathology, cholecystectomy or for diagnostic procedures to rule out intra-abdominal pathology
  Interventions: Other: Age-appropriate Wechsler Intelligence Test; Other: Disruptive Behavior Disorders Rating Scale; Other: Social Responsiveness Scale
- No Prenatal Anaesthesia Exposure: Children not exposed to general anaesthesia for non-obstetric or obstetric (e.g. cesarean section) surgery in utero
  Interventions: Other: Age-appropriate Wechsler Intelligence Test; Other: Disruptive Behavior Disorders Rating Scale; Other: Social Responsiveness Scale
- Prenatal exposure to maternal inflammation: Children prenatally exposed to maternal inflammation, specifically those born to mothers with inflammatory bowel disease (IBD)
  Interventions: Other: Age-appropriate Wechsler Intelligence Test; Other: Disruptive Behavior Disorders Rating Scale; Other: Social Responsiveness Scale

INTERVENTIONS:
Other: Age-appropriate Wechsler Intelligence Test — 2.5-6 years: Wechsler Preschool and Primary Scale of Intelligence for children (WPPSI IV)
  7-16 years: Wechsler Intelligence Scale for Children (WISC V)
  >17 years: Wechsler Adult Intelligence Scale (WAIS IV)
Other: Disruptive Behavior Disorders Rating Scale — Dutch version of the Disruptive Behavior Disorders Rating Scale
Other: Social Responsiveness Scale — 3-18 years: social responsiveness scale 2 (SRS-2)
  >19 years: Social Responsiveness Scale - Adult version (SRS-A)

SUMMARY:
Every year in the European Union, thousands of babies are exposed to anaesthesia before they are born because their mothers need surgery during pregnancy. While these surgeries are necessary, there is a concern that the anaesthesia might affect the baby's brain development. However, there isn't enough research to know for sure how this exposure might impact the child's intelligence or behavior later in life.

The goal of this cohort study is to compare the intelligence and neurodevelopmental outcome of children prenatally exposed to general anaesthesia for maternal abdominal surgery with those of unexposed children and with those of children prenatally exposed to maternal inflammation.

ELIGIBILITY:
Prenatal anaesthesia exposure:

Inclusion Criteria:

* Prenatal anaesthesia exposure: Children exposed in utero to maternal general anaesthesia to allow laparoscopy or laparotomy for appendicectomy, adnexal pathology, cholecystectomy or for diagnostic procedures to rule out intra-abdominal pathology
* No prenatal anaesthesia exposure: Children not exposed to general anaesthesia for non-obstetric or obstetric (e.g. cesarean section) surgery in utero
* Children exposed to inflammation: Children born to mothers diagnosed with inflammatory bowel disease (IBD) who had a flare-up during pregnancy without being exposed to general anaesthesia for non-obstetric or obstetric (e.g. cesarean section) surgery in utero.
* Children born in 2000-2023
* (Parental) informed consent

Exclusion Criteria:

* Children whose mothers underwent obstetric surgery or foetal surgery/interventions during the same pregnancy.
* No Dutch-speaking children
* Diagnosis of severe disability of genetic origin (e.g., Fragil X, Down syndrome,…), history of head trauma, major congenital birth defects

Ages: 2 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children from women who delivered in one of the participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Wechsler full-scale intelligence quotient | 1,5 hours (duration of intelligence testing and completion of questionnaires)
  Primary outcome will be the Wechsler full-scale intelligence quotient which will be assessed using the Wechsler Preschool and Primary Scale of Intelligence for children with an age of 2.5-6 years, the Wechsler Intelligence Scale for Children for children with an age of 7-16 years and the Wechsler Adult Intelligence Scale for children with an age of ≥ 17 years.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Devroe, MD, Phd, Principal Investigator — UZ Leuven
Locations (3):
- Belgium (3):
  - Imeldaziekenhuis, Bonheiden, Antwerpen
  - UZ Leuven, Leuven, Vlaams-Brabant
  - AZ Delta, Roeselare, West-Flanders

IPD SHARING:
Plan to Share IPD: No